CLINICAL TRIAL: NCT03606421
Title: Use of Novel MRI Techniques Before and After Brain Radiotherapy With Parallel Assessments of Neurocognitive Function
Brief Title: CBF and NCF Changes With Brain Radiation
Status: Recruiting | Type: Observational
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Other Study IDs: 18-5106
Record Dates: First submitted 2018-06-27; First posted 2018-07-30 (Actual); Last update posted 2024-06-18 (Actual); Status verified 2024-06

CONDITIONS: Neurocognitive Dysfunction; Brain Metastases
MeSH Terms: conditions — Cognition Disorders; Brain Neoplasms | interventions — Spermine Synthase

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Arm A: Patients in Arm A will be treated with stereotactic radiosurgery (SRS) which is a modern method of treating brain lesions that delivers a high amount of radiation to a small volume of the brain affected by a tumour; and is the standard of care for patients with a limited number of brain metastases.
  Interventions: Radiation: SRS and neurocognitive assessments
- Arm B.: Patients in Arm B will be treated with whole brain radiotherapy, due to the number of lesions in their brain.
  Interventions: Radiation: WBRT and neurocognitive assessments

INTERVENTIONS:
Radiation: SRS and neurocognitive assessments — Patients will be assessed for cerebral blood flow and their neurocognitive function based on a series of neurocognitive tests and questionnaires.
  Groups: Arm A
Radiation: WBRT and neurocognitive assessments — Patients will be assessed for cerebral blood flow and their neurocognitive function based on a series of neurocognitive tests and questionnaires.
  Groups: Arm B.

SUMMARY:
This study will be a dual-arm prospective longitudinal cohort study for patients with brain metastases, at least one of which is appropriate for radiotherapy, to explore brain and cognitive changes following SRS or WBRT and evaluate the feasibility of a novel MRI protocol to identify potential radiological biomarkers of NCF decline.

Patients diagnosed with brain mets will be assigned to either Arm A or Arm B, depending on their treatment plan. Patients in Arm A will be treated with SRS. Patients in Arm B will be treated with WBRT.

Patients' neurocognitive function will be assessed before their radiation treatment and followed up for 2 years post treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients with brain metastases will be included in this study. Patients with known malignancies but without brain metastases, or patients with primary brain tumors are not eligible for enrollment.
* MRI confirmed 1-10 lesions. Each lesion must not be intended for resection.
* No prior radiation therapy for brain tumours.
* For patients enrolled to arm B, ability to tolerate RespirAct. Based on studies in patients with severe cerebrovascular disease, an 8 - 16% drop-out rate at the time of the first exposure to RespirAct CVR testing is expected [9]. The fourth generation of this device has been associated with increased tolerability secondary to elimination of a physical rebreathing circuit replaced by a digital re-breath analog. This improvement is expected to achieve a drop-out rate significantly below 10%.
* Patients must have a GPA greater than or equal to 1.0.
* Patients must be able to provide informed consent. Patient consent must be appropriately obtained in accordance with applicable local and regulatory requirements. Each patient must sign a consent form prior to enrollment in the trial to document their willingness to participate.
* Patients must have sufficient fluency in English and sufficient motor and visual functioning (corrected or assisted as required) to complete the NCF-A battery.
* Patients must be accessible for treatment, AE assessment and follow- up.
* Limit to KPS ≥ 70 for patients in arm B; no limit for arm A
* Women/men of childbearing potential must have agreed to use a highly effective contraceptive. Women of childbearing potential will have a pregnancy test to determine eligibility.

Exclusion Criteria:

* Treatment plan respecting normal tissue tolerances using dose fractionation specified within the protocol cannot be achieved.
* Pregnant patients will be excluded from this study.
* Prior cranial radiotherapy
* Inability to complete MRI with contrast of the head, or a known allergy to gadolinium
* Metastatic germ cell tumor, small cell carcinoma, or lymphoma or any primary brain tumor.
* Patients with known malignancies but without brain metastases.
* Image Findings

  * Widespread definitive leptomeningeal metastasis
  * A brain metastasis that is located ≤ 2 mm of the optic chiasm
  * Evidence of midline shift
  * Fourth ventricular narrowing, concerning for hydrocephalus
* Patients who have undergone surgical resection of brain tumor are not eligible for enrollment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with brain metastases, at least one of which is appropriate for radiotherapy
Sampling Method: Non-Probability Sample
Enrollment: 110 (Estimated)
Dates: Start 2018-10-01 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
change in neurocognitive function (NCF) | Over 24 months
  To characterize change in NCF from baseline (pre-SRS treatment), to 24 months following using the NCF-A Battery

SECONDARY OUTCOMES:
Symptomatic Radiation Toxicity | 3-24 months
  A diagnosis of symptomatic radiation toxicity will be based on a clinical onset of symptoms and radiological findings of radionecrosis at 3-24 months following radiosurgery, with or without pathological confirmation
Local Failure | up to 24 months
  Local failure will be defined as one of the following (follow-up MRI or CT brain scans will be compared to the prior MRI or CT brain scan): Increase of > 25% in the size of any lesion or a new, non- contiguous lesion developed outside the radiosurgical bed (in the brain or meninges). Radionecrosis will not be considered tumor progression.
Distant Failure | up to 24 months
  Distant disease is considered to be new metastatic lesions in the brain or outside the brain following WBRT and SRS.
Survival | up to 24 months
  Survival time will be measured from the date the patient is enrolled in this study to death, due to any cause

CONTACTS AND LOCATIONS:
Locations (1):
- University Health Network, Toronto, Ontario, Canada